CLINICAL TRIAL: NCT03728140
Title: Can Embryo Transfer With Self-spent Culture Medium Improve Clinical Pregnancy Outcomes in Vitro Fertilization - Embryo Transfer Process?
Brief Title: Embryo Transfer With Self-spent Culture Medium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bin Wu (Other)
Responsible Party: Sponsor-Investigator, Bin Wu, Reproductive medcine, Jinan Central Hospital
Organization: Jinan Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: JianCH-RM001
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-12

CONDITIONS: in Vitro Fertilization
Keywords: Embryo Transfer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-spent Culture Medium (Experimental): Changing embryo transfer solution with self-spent culture medium
  Interventions: Procedure: Self-spent Culture Medium
- New Culture Medium (No Intervention): embryo transfer with new culture medium in IVF-ET

INTERVENTIONS:
Procedure: Self-spent Culture Medium — Replace embryo transfer solution with Self-spent culture medium in IVF-ET.
  Arms: Self-spent Culture Medium

SUMMARY:
Embryo Transfer With Self-spent Culture Medium or new Culture Medium in Vitro Fertilization - Embryo Transfer Process, to analyze which way can improve clinical pregnancy outcomes, is there a significant difference between the two?

DETAILED DESCRIPTION:
Although some metabolites are present in self-spent culture medium, there are some embryonic exocrine factors secreted by embryo.These factors may have a positive impact on embryo implantation and subsequent development. So it is necessary to compare the two ways of embryo transfer with Self-spent Culture Medium or New Culture Medium in vitro fertilization - embryo transfer process.

The purpose of this study is to analyze which way can improve clinical pregnancy and birth outcomes, is there a significant difference between the two?

ELIGIBILITY:
Inclusion Criteria:

* Infertility female patients with tubal factors,
* Infertile female patients with spouse factors

Exclusion Criteria:

* Intrauterine adhesions,
* Endometriosis,
* Primary ovarian insufficiency，
* Infectious disease

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in childbearing age intend to do IVF
Enrollment: 335 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yingchun zhang, Dr, Study Director — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-spent Culture Medium | New Culture Medium
Started | 160 (embryo transfer with self-spent culture medium) | 175 (embryo transfer with new culture medium)
Completed | 150 | 168
Not Completed | 10 | 7
Not completed — Abnormal embryo transfer operation | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-spent Culture Medium | New Culture Medium | Total
Number analyzed (Participants) | 150 | 168 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.31 (4.08) | 29.72 (4.77) | 29.99 (4.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 168 | 318
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 150 | 168 | 318
duration of infertility [Mean (Standard Deviation); unit: years] | 3.44 (2.24) | 3.58 (3.39) | 3.51 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Pregnant After 4 Weeks
Description: Observe the clinical pregnancy rate under different embryo transfer methods
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Self-spent Culture Medium | New Culture Medium
Number analyzed (Participants) | 150 | 168
Participants | 85 | 82

2. Primary Outcome: Live Birth
Description: Observe the live birth rate under different embryo transfer methods
Time Frame: 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Self-spent Culture Medium | New Culture Medium
Number analyzed (Participants) | 150 | 168
Participants | 78 | 74

ADVERSE EVENTS:
Time Frame: 1 year
Description: No any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research,
Groups:
- Self-spent Culture Medium: embryo transfer with self-spent culture medium
- New Culture Medium: embryo transfer with new culture medium
Arm/Group | Self-spent Culture Medium | New Culture Medium
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/168
Other Adverse Events (participants affected / at risk) | 0/150 | 0/168

LIMITATIONS AND CAVEATS:
Studies of larger sample sizes and studies on some other variables were needed to be further performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03728140/Prot_SAP_000.pdf